CLINICAL TRIAL: NCT05548426
Title: Pilot Study of Linezolid for Early Syphilis Treatment
Brief Title: Linezolid for Syphilis Pilot Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Universidad Peruana Cayetano Heredia (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jeffrey D Klausner, Clinical Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APP-22-04165
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Syphilis
Keywords: Linezolid; Treponema pallidum; Penicillin; Early Syphilis
MeSH Terms: conditions — Syphilis; Treponemal Infections | interventions — Linezolid; Penicillins; Penicillin G Benzathine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Linezolid 10 Day (Experimental): Oral linezolid 600mg, taken twice a day for 10 days
  Interventions: Drug: Group B, Linezolid 10d
- Benzathine Penicillin G (Active Comparator): Single intramuscular injection of 2.4 million units of benzathine penicillin G
  Interventions: Drug: Group A, Penicillin

INTERVENTIONS:
Drug: Group B, Linezolid 10d — Oral Linezolid 600mg, taken twice a day for 10 days
  Other Names: zyvox
  Arms: Linezolid 10 Day
Drug: Group A, Penicillin — Standard of care benzathine penicillin G, one intramuscular injection, 2.4MU
  Other Names: bicillin
  Arms: Benzathine Penicillin G

SUMMARY:
The study aims to evaluate the efficacy of linezolid for the treatment of syphilis.

DETAILED DESCRIPTION:
This will be a randomized, open-label, non-comparative, adaptive pilot trial to evaluate the efficacy of linezolid 600mg orally, twice a day, for five or ten days, using a contemporaneous historical control group benzathine penicillin G (single dose of 2.4 million units) in participants with and without HIV infection.

In total, 24 participants will be enrolled across multiple clinical sites in the United States. Participants will participate in follow-ups to monitor clinical outcomes and serological response (RPR titer) at 1 month, 3 months, and 6 months.

Study findings may identify an efficacious alternative syphilis treatment to penicillin that is effective for people living with HIV. Study findings may also help address the crisis of penicillin shortages, difficulty in administration, and offer options for those with penicillin allergy.

ELIGIBILITY:
Inclusion Criteria:

* 16 years of age or older
* Diagnosed cases of primary, secondary, or early latent syphilis with RPR titer ≥1:8 within 3 weeks prior to enrollment
* Able to provide informed consent
* For PLHIV: on treatment for HIV-infection and most recent viral load <200 copies/mL or most recent CD4 T-cell count >350 cells/mL

Exclusion Criteria:

* Pregnancy or a positive pregnancy test on the day of enrollment
* Participants who receive certain psychotropic medications, e.g., MAO inhibitors, SNRIs, SSRIs
* Patients showing signs and symptoms of neurosyphilis
* Serofast RPR titer
* Recent (<7 days) or concomitant antimicrobial therapy with azithromycin, doxycycline, ceftriaxone, cefixime, or other beta lactam antibiotics (e.g. amoxicillin)
* Linezolid or penicillin allergy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Response to Treatment | 6 months
  Percentage of linezolid participants with a 4-fold decrease or greater in the serum RPR titer by 180 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D Klausner, MD MPH, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Howard Brown Health, Chicago, Illinois
  - Open Arms HealthCare Center, Jackson, Mississippi

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers